CLINICAL TRIAL: NCT03970473
Title: Pulmonary Recruitment Maneuver With 15 or 30 cmH2O Pressure in Semi-Fowler Position: Which Provides Less Postoperative Shoulder Pain Following Gynecologic Laparoscopic Surgery
Brief Title: Pulmonary Recruitment Maneuver With 15 and 30 cmH2O Pressure to Reduce the Postoperative Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gulseren Yilmaz, Principal Investigator, M.D., Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Gulseren3
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Surgery
Keywords: gynecologic laparoscopic surgery; post-laparoscopic shoulder pain; pulmonary recruitment manoeuvre

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRM 30 cm H2O (Active Comparator): In this group, following the laparoscopic surgery and just before the extubation, patients will receive PRM with 30 cm H2O in the semi-fowler position.
  Interventions: Other: Pulmonary recruitment maneuver (PRM)- 30 cm H2O
- PRM 15 cm H2O (Active Comparator): In this group, following the laparoscopic surgery and just before the extubation, patients will receive PRM with 15 cm H2O in the semi-fowler position.
  Interventions: Other: Pulmonary recruitment maneuver (PRM)- 15 cm H2O

INTERVENTIONS:
Other: Pulmonary recruitment maneuver (PRM)- 30 cm H2O — Pulmonary recruitment maneuver (PRM) consists of five manual pulmonary inflations where each positive pressure inflation will be performed for 5 s at a maximum pressure of 30 cm H2O in the semi-fowler position (30° head-of-bed elevation ). PRM is performed after LS when the main umbilical port is remaining and aims to remove the remaining gas following LS.
  Arms: PRM 30 cm H2O
Other: Pulmonary recruitment maneuver (PRM)- 15 cm H2O — Pulmonary recruitment maneuver (PRM) consists of five manual pulmonary inflations where each positive pressure inflation will be performed for 5 s at a maximum pressure of 15 cm H2O in the semi-fowler position (30° head-of-bed elevation ). PRM is performed after LS when the main umbilical port is remaining and aims to remove the remaining gas following LS.
  Arms: PRM 15 cm H2O

SUMMARY:
Pulmonary recruitment maneuver (PRM) has been shown to reduce postoperative shoulder pain by removing excessive intraabdominal gas following laparoscopic surgery(LS). A recent study demonstrated that compared to PRM in the supine position, PRM at semi-fowler position provides better evacuation of the remaining intraabdominal gas following gynecologic LS.

This study aimed to compare the impact of PRM with 15 cm H2O and PRM with 30 cm H2O on postoperative shoulder pain in patients undergoing gynecologic LS.

DETAILED DESCRIPTION:
Pulmonary recruitment maneuver (PRM) consists of five manual pulmonary inflations where each positive pressure inflation was done for 5 s at a maximum pressure of 30-40 cm H2O in the neutral position. When used after laparoscopic surgery and just before the extubation, PRM has been shown to facilitate the removal of intraabdominal gas and thus reduce the postoperative shoulder pain which is associated with the volume of the gas accumulating under the diaphragm. A recent study demonstrated that compared to PRM in the supine position, PRM at semi-fowler position provides better evacuation of the remaining intraabdominal gas and less postoperative shoulder pain following gynecologic LS. However, whether a PRM with lower pressure is also effective in reducing postoperative intraabdominal gas and postoperative shoulder pain is of question. This study aimed to compare the impact of PRM with two pressures (15 cm H2O or 30 cm H2O) in addition to the semi-fowler position on postoperative shoulder pain in patients undergoing gynecologic LS.

ELIGIBILITY:
Inclusion Criteria:

* Must be scheduled for LS for benign causes
* Must be American Society of Anesthesiologists (ASA) class I or II.

Exclusion Criteria:

* Previous lung surgery
* Preexisting Emphysema
* Previous Pneumothorax

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Postoperative shoulder pain using a Visual Analogue Scale (VAS) based on a 0-10 scale, with 0 meaning no pain and 10 the most intense pain ever experienced | At postoperative 6, 12 and 24 hours using a visual analogue scale (VAS) based on a 0-10 scale, with 0 meaning no pain and 10 the most intense pain ever experienced.
  Change in postoperative shoulder pain between the two PRM pressure groups

CONTACTS AND LOCATIONS:
Overall Officials: Gulseren Yilmaz, MD, Principal Investigator — Kanuni Sultan Suleyman Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No